CLINICAL TRIAL: NCT07241975
Title: Real-world Experience With the Available Outpatient COVID-19 Therapies in Patients With Cancer: an Ambispective Cohort Study
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Angioletta Lasagna, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: CO_TER
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-02

CONDITIONS: Cancer Patients in Treatment Active Who Receive Early Out-patient Therapy Against SARS-CoV-2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The real-life efficacy of early antiviral therapies in cancer patients with COVID-19 is largely uncharacterized. From these unresolved issues, it is therefore necessary to fill these knowledge gaps by assessing the efficacy and safety of these therapies in combination with anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years diagnosed with and/or treated for solid tumors at the department of Oncologia of the Fondazione IRCCS Policlinico San Matteo
2. Prospective patients (or their or legal guardians) who have the ability to understand and be willing to sign a written informed consent document
3. Retrospective patients who have signed the institutional document allowing the use of their data for research on their disease

Exclusion Criteria:

* Patients who are unable to understand informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumors on active treatment who have COVID-19 infection and receive an early therapy are eligible.
  Patients admitted from January 2022 to December 2023 are candidate for the study. At the closure of the enrollment, we plan a further follow-up of 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
evaluate the rate of hospitalization for COVID-19 disease within 14 days in the patients with cancer using COVID-19 early therapies as per indication. | Data will be collected at T0 = start of COVID-19 therapy T1 = seven days after T0 T2 = 2 weeks after T0 T3 = one month after T0 T4 = + 3 months after T0 T5 = + 6 months after T0 T6 = + 12 months after T0

SECONDARY OUTCOMES:
To evaluate the mortality rate for COVID-19 disease | Data will be collected at T0 = start of COVID-19 therapy T1 = seven days after T0 T2 = 2 weeks after T0 T3 = one month after T0 T4 = + 3 months after T0 T5 = + 6 months after T0 T6 = + 12 months after T0
To evaluate the time to COVID 19 symptoms resolution | Data will be collected at T0 = start of COVID-19 therapy T1 = seven days after T0 T2 = 2 weeks after T0 T3 = one month after T0 T4 = + 3 months after T0 T5 = + 6 months after T0 T6 = + 12 months after T0
To evaluate the time to nasal swab viral clearance | Data will be collected at T0 = start of COVID-19 therapy T1 = seven days after T0 T2 = 2 weeks after T0 T3 = one month after T0 T4 = + 3 months after T0 T5 = + 6 months after T0 T6 = + 12 months after T0
To evaluate the time of the re-start of the oncological treatment | Data will be collected at T0 = start of COVID-19 therapy T1 = seven days after T0 T2 = 2 weeks after T0 T3 = one month after T0 T4 = + 3 months after T0 T5 = + 6 months after T0 T6 = + 12 months after T0
To evaluate the incidence of drug-related adverse events | Data will be collected at T0 = start of COVID-19 therapy T1 = seven days after T0 T2 = 2 weeks after T0 T3 = one month after T0 T4 = + 3 months after T0 T5 = + 6 months after T0 T6 = + 12 months after T0
To evaluate the incidence of long COVID symptoms according to WHO case definition | Data will be collected at T0 = start of COVID-19 therapy T1 = seven days after T0 T2 = 2 weeks after T0 T3 = one month after T0 T4 = + 3 months after T0 T5 = + 6 months after T0 T6 = + 12 months after T0

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Oncologia, Pavia, Pavia, Italy